CLINICAL TRIAL: NCT06690541
Title: A Real-world Study to Explore Therapeutic Changing Mode of Locally Therapy During 1L Lorlatinib Treatment in Unresectable ALK+ NSCLC Patients
Brief Title: Real-world Study of Local Therapy Changes During 1L Lorlatinib in Unresectable ALK+ NSCLC
Acronym: COMLORLA
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Zhao, Deputy Director of Thoracic Cancer Center;, Peking University Cancer Hospital & Institute
Other Study IDs: 2024YJZ112
Record Dates: First submitted 2024-11-07; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer, Non-Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Lorlatinib 100 mg — Patients received continuous daily PO dosing of lorlatinib 100mg QD from the date of first dosing (per the current protocol) or until one of the following criteria were met (whichever occurred first): disease progression; initiation of a new anticancer therapy; unacceptable toxicities; global deterioration of health-related symptoms; pregnancy; withdrawal of consent; loss to follow-up; death; investigator decision dictated by protocol non-compliance; or study termination.

SUMMARY:
This real-word study is designed to prospectively explore whether local treatment (surgery, ablation, radiotherapy and others) can prolong the time to treatment discontinuation during 1L lorlatinib treatment in Chinese patients with unresectable ALK+ NSCLC. Participation in this study is not intended to change the routine treatment received as determined by their attending physicians. Patients will be treated according to the routine medical practice in terms of visit frequency and types of assessments performed.

ELIGIBILITY:
1 Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1.1. Diagnosis:

1. Study Population: Patients with histologically or cytologically confirmed diagnosis of locally advanced [(Stage IIIB/C not amenable for multimodality treatment) or metastatic (Stage IV) by American Joint Committee on Cancer (AJCC) v 7.0] ALK-positive NSCLC where ALK status is determined by the Ventana ALK (D5F3) Companion Diagnostic (CDx) IHC test performed on the Ventana ULTRA or XT Platforms, FISH, PCR, or next generation sequencing (NGS), or circulating tumor DNA (ctDNA).
2. Tumor Requirements: At least 1 measurable target lesion per RECIST v. 1.1 that has not been previously irradiated. Brain metastases are allowed.

1.2. No prior systemic treatment for advanced (Stage IIIB/C not amenable for multimodality treatment) or metastatic (Stage IV) disease.

1.3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0, 1, 2 or 3.

1.4. Age ≥18 years. 1.5. Adequate Liver Function, including:

1. Total serum bilirubin ≤1.5 x ULN;
2. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN (≤5.0 x ULN in case of liver metastases).

1.6. Life expectancy at least 6 months. 1.7. Serum pregnancy test (for females of childbearing potential) negative at screening. Female patients of non-childbearing potential must meet at least 1 of the following criteria:

1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause (which may be confirmed with a serum follicle-stimulating hormone [FSH] level confirming the postmenopausal state if appropriate);
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential. 1.8. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

1.9. Willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures. 2.Exclusion Criteria

Subjects presenting with any of the following characteristics/conditions will not be included in this clinical study:

2.1. Major surgery within 4 weeks prior to randomization. Minor surgical procedures (e.g., port insertion) are not excluded, but sufficient time should have passed for adequate wound healing.

2.2. Radiation therapy within 2 weeks prior to enrollment, including stereotactic or partial brain irradiation. Patients who complete whole brain irradiation within 4 weeks prior to randomization or palliative radiation therapy outside of the CNS within 48 hours prior to randomization will also not be included in the study.

2.3. Gastrointestinal abnormalities, including inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection or lap band; active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease; treatment for active peptic ulcer disease in the past 6 months; malabsorption syndromes.

2.4. Known prior or suspected severe hypersensitivity to study drugs or any component in their formulations.

2.5. History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis.

2.6. Evidence of active malignancy (other than NSCLC, non-melanoma skin cancer, or localized prostate cancer or any in situ cancer which does not currently require treatment) within the last 3 years prior to randomization.

2.7. Concurrent use of any of the following food or drugs (consult the sponsor if in doubt whether a food or a drug fall into any of the above categories) within 12 days prior to the first dose of lorlatinib.

1. Known strong CYP3A inhibitors (e.g., strong CYP3A inhibitors: grapefruit juice or grapefruit/grapefruit related citrus fruits [eg, Seville oranges, pomelos], boceprevir, cobicistat, conivaptan, itraconazole, ketoconazole, posaconazole, ritonavir alone and with danoprevir or elvitegravir or indinavir or lopinavir or paritaprevir or ombitasvir or dasabuvir or saquinavir or tipranavir, telaprevir, troleandomycin, and voriconazole. The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
2. Known CYP3A substrates with narrow therapeutic index, such as astemizole*, terfenadine*, cisapride*, pimozide, quinidine, tacrolimus, cyclosporine, sirolimus, alfentanil, fentanyl (including transdermal patch) or ergot alkaloids (ergotamine, dihydroergotamine) (*withdrawn from US market).
3. Known strong CYP3A inducers (e.g., carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's Wort). d. Known P-gp substrates with a narrow therapeutic index (e.g., digoxin).

2.8. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

2.9. Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed diagnosis of locally advanced [(Stage IIIB/C not amenable for multimodality treatment) or metastatic (Stage IV) by American Joint Committee on Cancer (AJCC) v 7.0] ALK-positive NSCLC where ALK status is determined by the Ventana ALK (D5F3) Companion Diagnostic (CDx) IHC test performed on the Ventana ULTRA or XT Platforms, FISH, PCR, or next generation sequencing (NGS), or circulating tumor DNA (ctDNA).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Time-to treatment discontinuation (TTD) | From November 2024 to April 2027
  Time-to treatment discontinuation is defined as the time from start of treatment to the date of discontinuation of these therapeutic methods.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From November 2024 to April 2027
  proportion of patients with a Complete Response (CR) or Partial Response (PR) as a best response during the lorlatinib treatment. Responses to treatment will be defined according to investigator
Duration of response (DOR) | From November 2024 to April 2027
  time between the first documentation of objective response and the first documentation of disease progression or death from any cause whichever occurred first, for participants with a confirmed objective response of CR or PR.
Time to Progression (TTP) | From November 2024 to April 2027
  Based on Investigator's Assessment
Intracranial Objective Response Rate (IC-ORR) | From November 2024 to April 2027
  proportion of patients with intracranial objective response of complete response (CR) or partial response (PR) as a best response in the subset of patients with at least 1 intracranial lesion assessed by investigator.
Intracranial Time to Progression (IC-TTP) | From November 2024 to April 2027
  Time from inclusion to the date of the first documentation of disease progression of intracranial disease, based on either new brain metastases or progression of existing brain metastases.
Overall Survival (OS) | From November 2024 to April 2027
  Time from inclusion to date of death from any cause.
Safety: To explore the adverse events (AEs), the dose modification and the reason for interruption or discontinuation of lorlatinib in first line for Chinese patients with ALK-positive locally advanced or metastatic NSCLC recorded in medical records | From November 2024 to April 2027
Proportion of patients experiencing a 10-points change from baseline in total score for the EORTC QLQ-C30 | From November 2024 to April 2027
  evaluate Health-related Quality of life (HRQoL) of ALK- positive locally advanced or metastatic NSCLC patients treated with lorlatinib in first-line using the EORTC QLQ-C30 questionnaires
Dynamic molecular response | From November 2024 to April 2027
  Mutational Analysis; measured by next-generation sequencing (NGS) if available in real world setting;
Safety and tolerability of the therapeutic changing mode | From November 2024 to April 2027
  Safety profile according to CTCAE v.5

OTHER OUTCOMES:
Dynamic ctDNA change during lorlatinib treatment | From November 2024 to April 2027
  Plasma samples collected at several timepoints, analyzed by next-generation sequencing
Biomarkers of sensitivity or resistance to lorlatinib in no-prior ALK-TKIs treatment tumor tissue and peripheral blood if available in real world setting | From November 2024 to April 2027

DOCUMENTS (2):
  • Study Protocol (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT06690541/Prot_000.pdf
  • Informed Consent Form (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT06690541/ICF_001.pdf